CLINICAL TRIAL: NCT01590381
Title: Assessment of the Immune Status of New Health Care Workers in the Israel Defense Forces (IDF) Vaccinated in Infancy Against Hepatitis B Virus (HBV), Before and After a Booster Dose.
Brief Title: Assessment of HBV Vaccine Immunity After 18 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Other Study IDs: IDF 1047-2011
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Hepatitis b Vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples from study subjects vaccinated at infancy, before and after booster dose.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- personnel in medical training - COURSE 1
- personnel in medical training - COURSE 2
- personnel in medical training - COURSE 3
- personnel in medical training - COURSE 4
- personnel in medical training - COURSE 5
- personnel in medical training - COURSE 6
- personnel in medical training - COURSE 7
- personnel in medical training - COURSE 8
- personnel in medical training - COURSE 9
- personnel in medical training - COURSE 10

SUMMARY:
The purpose of this study is to assess HBV immunity and institute policy regarding the Hepatitis B vaccination practices in the IDF among a cohort that was vaccinated during infancy.

DETAILED DESCRIPTION:
The study population will consist of both males and females who were born after January 1st 1992, who are in medical training at the Medical Corps Training Base. Demographic information will be obtained through a questionnaire given to the soldiers in the study , as well as the IDF computerized personnel information database.

This study is designed to determine HBV vaccination policy among new HCWs in the IDF, who were vaccinated during infancy. This population was recruited to the IDF since the second half of 2010. Therefore, it is necessary to conduct this study on new HCWs that will be receiving the routine HBV vaccination and that will be at risk for HBV infection in the future due to their occupation in the army (HCWs, etc).

ELIGIBILITY:
Inclusion Criteria:

1. Soldiers born on or after January 1st, 1992
2. Soldiers taking part in a medical training course
3. Soldiers that signed an informed consent form

Exclusion Criteria:

1. Born before January 1st, 1992
2. Soldiers with previous known infection with HBV
3. Soldiers with documented evidence of immunity against HBV
4. Soldiers that refuse to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of both males and females who were born after January 1st 1992, who are in medical training at the Medical Corps Training Base.
Sampling Method: Probability Sample
Enrollment: 545 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hartal, MD, Principal Investigator — International Diabetes Federation
Locations (1):
- Israeli Defense Forces, Tel Aviv, Israel